CLINICAL TRIAL: NCT06993363
Title: Effect of Adding Kinesotaping to Quadriceps Strengthening on Knee Function in Patients With Osgood Schlatter
Brief Title: Kinesotaping and Strengthening Exercises in Treatment of Osgood-Schlatter Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Doaa Rafat, Assisstant professor of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005847
Record Dates: First submitted 2025-05-19; First posted 2025-05-28 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Osgood-Schlatter Disease
Keywords: Osgood-Schlatter disease; Knee function; kinesotaping; strengthening exercises
MeSH Terms: conditions — Osteochondrosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Patients will receive strengthening exercises to quadriceps muscle and stretching exercises to hamstring and calf muscles
  Interventions: Other: Quadriceps Strengthening; Other: Hamstring and calf stretching exercise
- Group B (Experimental): Patients will receive kinesotaping, strengthening exercises to quadriceps muscle and stretching exercises to hamstring and calf muscles
  Interventions: Other: Quadriceps Strengthening; Other: Hamstring and calf stretching exercise; Other: Kinesotaping application

INTERVENTIONS:
Other: Quadriceps Strengthening — Static Quad Pull the toes up towards your shin, push your knee into the bed to tighten the quad muscles. This should cause your heel to slightly lift off the bed. Hold for 7 seconds. Repeat on affected leg.
  Straight leg raising
  * Lie on back with hips square and legs laid out comfortably on the floor
  * Bend the knee of non-injured leg at a 90-degree angle, planting the foot flatly on the floor.
  * Stabilize the muscles on your straight leg by contracting your quadriceps (the group of muscles on the front of your thigh).
  * Inhaling slowly, lift the straight leg six inches off the ground.
  * Hold for three seconds.
  * Exhaling slowly, lower the leg to the floor with control
  * Relax and repeat 10 times more.
Other: Hamstring and calf stretching exercise — Hamstring stretching exercise will be done in the long sitting position. The patient will be instructed to keep his affected knee always extended while folding the other leg to the side then he will bend his trunk forward as much as he could in order to touch his toes by his fingers.
  Calf muscle stretching: The patient will be positioned in the long-sitting with the knees extended. The patient will be instructed to pull his foot into dorsiflexion as much as he could with the assistance of a rolled towel holding this position for 30 seconds (Fig14). The patient will then be instructed to go back to starting position and relax for 30 seconds. This exercise will be done 5 times per session.
Other: Kinesotaping application — 1 full 25cm strip of KT Tape cut in half. Apply one hour before beginning activity. Clean dirt, oils and lotions from area. After application rub tape vigorously to activate adhesive. Bend the knee at a 90 degree angle Anchor the middle of a half strip of tape diagonally over the point of pain with 80% stretch. Apply ends of tape without stretch.
  Anchor the middle of a second half strip across the first strip to form an X pattern over the point of pain with 80% stretch.
  Arms: Group B

SUMMARY:
The purpose of this study is to investigate the effect of adding kinesotaping to quadriceps strengthening exercises on muscle strength, pain, function and range of motion of knee joint in patients with Osgood-Schlatter disease (OSD).

DETAILED DESCRIPTION:
60 patients will be participated in this study. The patients of both genders with age ranges from 18 -25 years old. The sample will randomly be divided into two groups.

Group A: will receive strengthening exercise for quadriceps muscle and stretching exercises for hamstring and calf muscles Group B: will receive kinesoatping, strengthening exercises for quadriceps muscle and stretching exercises for hamstring and calf muscles .

All subject will receive the treatment for 6 weeks, All subjects will assign consent form before starting this study and will be explained the purpose of this study before any application.

Outcome measurements:

1. Quadriceps muscles strength will be assessed by hand held dynamotor.
2. Pain intensity will be measured by visual analog scale.
3. Disability function of knee will be measured by lower extremity functional scale (LEFS-Ar).
4. Range of motion of knee joint will be measured by smart phone application for range of motion measurement.

Data will be collected prior to first session as pre-test measure and at the end of last treatment session as post-test treatment.

ELIGIBILITY:
Inclusion Criteria:

1 - Age - 18 years to 25 years 2. Knee Osgood schlatter disease as per diagnosed by orthopaedisit 3. Duration of knee pain is 4-5 weeks during 6 months prior to study. 4- patients from both gender 5- BMI from 18 Kg/M2 to 25 Kg/M2

Exclusion Criteria:

1. History of low back pain.
2. Trauma to the knee joint.
3. Loss of joint play in tibiofemoral and patellofemoral articulations.
4. Lower extremity fracture and surgery.
5. Neurological deficit or movement disorder.
6. If they had meniscal symptoms.
7. If they had rheumatoid.
8. If they had osteoarthritis.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
Change in muscle strength | at first week and after 6 weeks of treatment
  Quadriceps muscle strength will be assessed by hand held dynamo-meter.

SECONDARY OUTCOMES:
Change in Pain level | at first week and after 6 weeks of treatment
  Pain threshold will be assessed by visual analogue scale
Change in functional disability | at first week and after 6 weeks of treatment
  Functional disability will assessed by lower extremity functional scale
Knee joint range of motion | at first week and after 6 weeks of treatment
  11. Knee range of motion (flexion, extension) will be assessed by smart phone application (Doctor Goniometer) for range of motion measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Neveen Abdelatif Professor of physical therapy - Cairo University, Professor, Study Chair — Department of Basic sciences for physical therapy, Faculty of Physical Therapy , Cairo university, Cairo, Egypt
Locations (1):
- Physical therapy College - Cairo university, Cairo, Egypt